

## **University Hospital of Pisa**

University Operative Emergency Surgery unit Director: Prof. M. Chiarugi

## PROJECT EXPERIMENTAL NON-PROFIT CLINICAL STUDY

Pisa, January 18<sup>th</sup>, 2017

Principal Investigator

Prof. Massimo Chiarugi

 ${\tt Co-Investigator}$ 

Dr. Dario Tartaglia

## Clinical Study Title

Laparoscopic peritoneal lavage versus laparoscopic sigmoidectomy in perforated Acute diverticulitis: A multicentric, prospective and observational study

NCT number: 03008707

## Statistical analysis

Continuous data were presented as mean  $\pm$  standard deviation unless indicated otherwise.

Qualitative data were expressed as frequency and percentage. The Student's t-test or Mann-Whitney U test, when data were not normally distributed, were used to perform a comparison of continuous quantitative data. Pearson's chi-square or Fisher's exact tests were comparing categorical qualitative variables, used appropriate. A p-value < 0.05 considered was statistically significant. All analyses were carried out using XLSTAT software (Addinsoft, NY, USA)